CLINICAL TRIAL: NCT02595320
Title: Randomized Open-label Trial of Dose Dense, Fixed Dose Capecitabine Compared to Standard Dose Capecitabine in Metastatic Breast Cancer and Advanced/Metastatic Gastrointestinal Cancers.
Brief Title: Capecitabine in Metastatic Breast and GI Cancers
Acronym: X7-7
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qamar Khan (Other)
Responsible Party: Sponsor-Investigator, Qamar Khan, Principal Investigator, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-IIT-X7-7
Record Dates: First submitted 2015-10-02; First posted 2015-11-03 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Gastrointestinal Cancer
Keywords: breast, gastrointestinal,capecitabine, cancer, metastatic
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): capecitabine, 1500 mg, twice a day for 7 days on then 7 days off
  Interventions: Drug: Capecitabine
- Group B (Active Comparator): capecitabine, 1250 mg/m2 OR 1000 mg/m2, twice a day for 14 days on then 7 days off
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be given to participants in Arm A at 1500 mg PO BID for 7 days, followed by a 7 day rest (7-7).
  Capecitabine will be given to participants in group B at 1250 mg/m2 OR 1000 mg/m2 PO BID for 14 days, followed by a 7 day rest (14-7).
  Other Names: Xeloda®

SUMMARY:
The purpose of this study is compare different doses of capecitabine to see if one is better than the other in terms of efficacy and toxicity.

DETAILED DESCRIPTION:
Goals of treatment of metastatic breast cancer remain largely comfort care. However, there has been improvement in median survival among women with metastatic disease over the last two decades, mainly due to availability of more effective agents. Women are now living longer with metastatic disease and are on therapy for longer periods of time. Therefore, it is increasingly important for effective therapies to be associated with less toxicity so that women can enjoy a better overall quality of life. Similar to breast cancer, goals of treatment of various GI malignancies (including metastatic colorectal cancer, metastatic gastric and esophageal cancers, and unresectable or metastatic pancreatic cancer and cholangiocarcinoma) are largely comfort care and it is important to minimize toxicity from therapy during the treatment for metastatic disease.

Capecitabine is a unique chemotherapeutic agent for two reasons. It is the only oral chemotherapy drug available to treat breast and GI malignancies, making it convenient for patients. In addition, whereas all other cytotoxic chemotherapy agents can be administered for only a few months at a time because of development of cumulative toxicities, capecitabine can be continued for many months to years if toxicities can be managed. However the optimal dosing schedule of capecitabine is not known.

This is the basis for the proposed randomized phase II trial, to compare the efficacy and tolerability of capecitabine 1500 milligrams (mg) twice a day (BID), 7 days on and 7 days off schedule to capecitabine 1250 milligrams/meters squared (mg/m2) BID, 14 days on and 7 days off) or 1000 mg/m2 BID, 14 days on and 7 days off, in women with metastatic breast cancer or patients with advanced/metastatic GI cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with metastatic breast cancer OR men and women with metastatic gastrointestinal (GI) cancer
* There is no limit to the number of prior chemotherapy or endocrine therapy regimens received. Use of a previous fluoropyrimidine-containing regimen in advanced / metastatic setting is permitted as long as the subject discontinued the regimen for reasons other than progression.
* No restriction on the use of fluoropyrimidine-containing regimen in the neoadjuvant or adjuvant setting
* For metastatic colorectal cancers, patients starting maintenance capecitabine after a course of oxaliplatin or irinotecan based chemotherapy are eligible.
* Measurable or non-measurable disease per RECIST criteria 1.1
* Must have completed prior chemotherapy or radiation therapy at least 2 weeks prior to registration
* Pathologic confirmation of respective malignancies. Biopsy of metastatic disease is preferred but not mandatory.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) Performance Score (PS) 0-2
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,000/ microLiter (uL)
  * hemoglobin ≥ 7 g/L
  * platelets ≥ 50,000/uL
  * total bilirubin ≤ 2 X the Institutional Upper Limit of Normal (IULN)
  * o Aspartate Aminotransferase (AST) ( Serum Glutamic Oxaloacetic Transaminase [SGOT]) ≤ 5 X IULN
  * Alanine Aminotransferase (ALT) (Serum Pyruvic Glutamic Transaminase [SPGT]) ≤ 5 X IULN
  * creatinine clearance > 50 milliliters per minute (ml/min)
* Women of childbearing potential must agree to use adequate contraception.
* Subjects may have previously treated brain or Central Nervous System (CNS) metastasis with radiation completed at least 2 weeks prior to registration. Prior radiation to places other than CNS disease must be completed at least 14 days prior to registration. Any number of prior radiation therapy regimens is allowed provided all toxicity of prior therapy is resolved to grade 1 or less.
* Life expectancy of >3 months

Exclusion Criteria:

* Patient has used Capecitabine in a past regimen for metastatic disease.
* Patient is currently using, or planning to use another investigational agent.
* Patient with known Dihydropyrimidine Dehydrogenase (DPD) deficiency
* Patient has symptomatic brain or CNS metastases.
* Patient has leptomeningeal disease
* Patient is pregnant or nursing
* Subjects must have no barriers to taking oral medications, for example uncontrolled nausea, vomiting, diarrhea at baseline, lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome.
* No recent (≤ 3months) of partial or complete bowel obstruction unless surgically corrected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Twelve-week Progression Free Survival (cohort 1 only) | 12 weeks from the date of registration into the study
  As the percentage of patients with progression from the date of registration to 12 weeks from that date

SECONDARY OUTCOMES:
Grade 3 or higher toxicity (cohorts 1 and 2) | From Day 1 of treatment, throughout treatment, up to 2 years from Day 1 of treatment
  Percentage of patients having grade 3 or higher toxicity from the date of first treatment dose during the trial therapy to patient develops Grade 3 or higher toxicity.

OTHER OUTCOMES:
Objective response rate (cohorts 1 and 2) | From Day 1 of treatment, throughout treatment, up to 2 years from Day 1 of treatment
  Objective response rate (complete and partial in subset of patients with measurable disease) from date of first treatment dose to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Qamar Khan, MD, Principal Investigator — University of Kansas Cancer Center - CRC
Locations (15):
- United States (15):
  - University of Kansas Cancer Center - CRC, Fairway, Kansas
  - St. Catherine Hospital - Central Care Cancer Center, Garden City, Kansas
  - Heartland Cancer Center - Central Care Cancer Center, Great Bend, Kansas
  - Hays Medical Center Dreiling-Schmidt Cancer Institute, Hays, Kansas
  - University of Kansas Cancer Center - West, Kansas City, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - Via Christi Cancer Center, Pittsburg, Kansas
  - Salina Regional Health, Salina, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - University of Kansas Cancer Center - Westwood, Westwood, Kansas
  - Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chia SK, Speers CH, D'yachkova Y, Kang A, Malfair-Taylor S, Barnett J, Coldman A, Gelmon KA, O'reilly SE, Olivotto IA. The impact of new chemotherapeutic and hormone agents on survival in a population-based cohort of women with metastatic breast cancer. Cancer. 2007 Sep 1;110(5):973-9. doi: 10.1002/cncr.22867. PMID 17647245
- [Background] Liu G, Franssen E, Fitch MI, Warner E. Patient preferences for oral versus intravenous palliative chemotherapy. J Clin Oncol. 1997 Jan;15(1):110-5. doi: 10.1200/JCO.1997.15.1.110. PMID 8996131
- [Background] Hofheinz RD, Wenz F, Post S, Matzdorff A, Laechelt S, Hartmann JT, Muller L, Link H, Moehler M, Kettner E, Fritz E, Hieber U, Lindemann HW, Grunewald M, Kremers S, Constantin C, Hipp M, Hartung G, Gencer D, Kienle P, Burkholder I, Hochhaus A. Chemoradiotherapy with capecitabine versus fluorouracil for locally advanced rectal cancer: a randomised, multicentre, non-inferiority, phase 3 trial. Lancet Oncol. 2012 Jun;13(6):579-88. doi: 10.1016/S1470-2045(12)70116-X. Epub 2012 Apr 13. PMID 22503032
- [Background] Kopf B, De Giorgi U, Zago S, Carminati O, Rosti G, Marangolo M. Innovative therapy for patients with brain metastases: oral treatments. J Chemother. 2004 Nov;16 Suppl 5:94-7. doi: 10.1080/1120009x.2004.11782396. PMID 15675490
- [Background] Fumoleau P, Largillier R, Clippe C, Dieras V, Orfeuvre H, Lesimple T, Culine S, Audhuy B, Serin D, Cure H, Vuillemin E, Morere JF, Montestruc F, Mouri Z, Namer M. Multicentre, phase II study evaluating capecitabine monotherapy in patients with anthracycline- and taxane-pretreated metastatic breast cancer. Eur J Cancer. 2004 Mar;40(4):536-42. doi: 10.1016/j.ejca.2003.11.007. PMID 14962720
- [Background] Oshaughnessy JA, Blum J, Moiseyenko V, Jones SE, Miles D, Bell D, Rosso R, Mauriac L, Osterwalder B, Burger HU, Laws S. Randomized, open-label, phase II trial of oral capecitabine (Xeloda) vs. a reference arm of intravenous CMF (cyclophosphamide, methotrexate and 5-fluorouracil) as first-line therapy for advanced/metastatic breast cancer. Ann Oncol. 2001 Sep;12(9):1247-54. doi: 10.1023/a:1012281104865. PMID 11697835
- [Background] Blum JL, Dieras V, Lo Russo PM, Horton J, Rutman O, Buzdar A, Osterwalder B. Multicenter, Phase II study of capecitabine in taxane-pretreated metastatic breast carcinoma patients. Cancer. 2001 Oct 1;92(7):1759-68. doi: 10.1002/1097-0142(20011001)92:73.0.co;2-a. PMID 11745247
- [Background] Blum JL, Jones SE, Buzdar AU, LoRusso PM, Kuter I, Vogel C, Osterwalder B, Burger HU, Brown CS, Griffin T. Multicenter phase II study of capecitabine in paclitaxel-refractory metastatic breast cancer. J Clin Oncol. 1999 Feb;17(2):485-93. doi: 10.1200/JCO.1999.17.2.485. PMID 10080589
- [Background] Mackean M, Planting A, Twelves C, Schellens J, Allman D, Osterwalder B, Reigner B, Griffin T, Kaye S, Verweij J. Phase I and pharmacologic study of intermittent twice-daily oral therapy with capecitabine in patients with advanced and/or metastatic cancer. J Clin Oncol. 1998 Sep;16(9):2977-85. doi: 10.1200/JCO.1998.16.9.2977. PMID 9738566
- [Background] Leonard R, O'Shaughnessy J, Vukelja S, Gorbounova V, Chan-Navarro CA, Maraninchi D, Barak-Wigler N, McKendrick JJ, Harker WG, Bexon AS, Twelves C. Detailed analysis of a randomized phase III trial: can the tolerability of capecitabine plus docetaxel be improved without compromising its survival advantage? Ann Oncol. 2006 Sep;17(9):1379-85. doi: 10.1093/annonc/mdl134. PMID 16966367
- [Background] Norton L. Conceptual and practical implications of breast tissue geometry: toward a more effective, less toxic therapy. Oncologist. 2005 Jun-Jul;10(6):370-81. doi: 10.1634/theoncologist.10-6-370. PMID 15967831
- [Background] Traina TA, Dugan U, Higgins B, Kolinsky K, Theodoulou M, Hudis CA, Norton L. Optimizing chemotherapy dose and schedule by Norton-Simon mathematical modeling. Breast Dis. 2010;31(1):7-18. doi: 10.3233/BD-2009-0290. PMID 20519801
- [Background] Traina TA, Theodoulou M, Feigin K, Patil S, Tan KL, Edwards C, Dugan U, Norton L, Hudis C. Phase I study of a novel capecitabine schedule based on the Norton-Simon mathematical model in patients with metastatic breast cancer. J Clin Oncol. 2008 Apr 10;26(11):1797-802. doi: 10.1200/JCO.2007.13.8388. PMID 18398145
- [Background] Gajria D, Feigin K, Tan LK, Patil S, Geneus S, Theodoulou M, Norton L, Hudis CA, Traina TA. Phase 2 trial of a novel capecitabine dosing schedule in combination with bevacizumab for patients with metastatic breast cancer. Cancer. 2011 Sep 15;117(18):4125-31. doi: 10.1002/cncr.25992. Epub 2011 Mar 8. PMID 21387266
- [Background] Ou SH, Holcombe RF. Capecitabine in advanced gastric or oesophagogastric cancer: a viewpoint by Sai-Hong Ignatius Ou and Randall F. Holcombe. Drugs. 2007;67(4):611-2. doi: 10.2165/00003495-200767040-00011. No abstract available. PMID 17352521
- [Background] Evans TR, Pentheroudakis G, Paul J, McInnes A, Blackie R, Raby N, Morrison R, Fullarton GM, Soukop M, McDonald AC. A phase I and pharmacokinetic study of capecitabine in combination with epirubicin and cisplatin in patients with inoperable oesophago-gastric adenocarcinoma. Ann Oncol. 2002 Sep;13(9):1469-78. doi: 10.1093/annonc/mdf243. PMID 12196374
- [Background] Hong YS, Song SY, Lee SI, Chung HC, Choi SH, Noh SH, Park JN, Han JY, Kang JH, Lee KS, Cho JY. A phase II trial of capecitabine in previously untreated patients with advanced and/or metastatic gastric cancer. Ann Oncol. 2004 Sep;15(9):1344-7. doi: 10.1093/annonc/mdh343. PMID 15319239
- [Background] Koizumi W, Saigenji K, Ujiie S, Terashima M, Sakata Y, Taguchi T; Clinical Study Group of Capecitabine. A pilot phase II study of capecitabine in advanced or recurrent gastric cancer. Oncology. 2003;64(3):232-6. doi: 10.1159/000069313. PMID 12697963
- [Background] Lee JL, Kang YK, Kang HJ, Lee KH, Zang DY, Ryoo BY, Kim JG, Park SR, Kang WK, Shin DB, Ryu MH, Chang HM, Kim TW, Baek JH, Min YJ. A randomised multicentre phase II trial of capecitabine vs S-1 as first-line treatment in elderly patients with metastatic or recurrent unresectable gastric cancer. Br J Cancer. 2008 Aug 19;99(4):584-90. doi: 10.1038/sj.bjc.6604536. Epub 2008 Jul 29. PMID 18665164
- [Background] Qiu MZ, Wei XL, Zhang DS, Jin Y, Zhou YX, Wang DS, Ren C, Bai L, Luo HY, Wang ZQ, Wang FH, Li YH, Yang DJ, Xu RH. Efficacy and safety of capecitabine as maintenance treatment after first-line chemotherapy using oxaliplatin and capecitabine in advanced gastric adenocarcinoma patients: a prospective observation. Tumour Biol. 2014 May;35(5):4369-75. doi: 10.1007/s13277-013-1574-5. Epub 2014 Feb 11. PMID 24515655
- [Background] Ajani J. Review of capecitabine as oral treatment of gastric, gastroesophageal, and esophageal cancers. Cancer. 2006 Jul 15;107(2):221-31. doi: 10.1002/cncr.21986. PMID 16770784
- [Background] Cartwright TH, Cohn A, Varkey JA, Chen YM, Szatrowski TP, Cox JV, Schulz JJ. Phase II study of oral capecitabine in patients with advanced or metastatic pancreatic cancer. J Clin Oncol. 2002 Jan 1;20(1):160-4. doi: 10.1200/JCO.2002.20.1.160. PMID 11773165
- [Background] Boeck S, Wilkowski R, Bruns CJ, Issels RD, Schulz C, Moosmann N, Laessig D, Haas M, Golf A, Heinemann V. Oral capecitabine in gemcitabine-pretreated patients with advanced pancreatic cancer. Oncology. 2007;73(3-4):221-7. doi: 10.1159/000127413. Epub 2008 Apr 17. PMID 18424886
- [Background] Saadati H, Saif MW. Capecitabine as salvage therapy for a pancreatic cancer patient with extensive liver metastases and associated impairment of liver function. JOP. 2008 May 8;9(3):354-6. No abstract available. PMID 18469454
- [Background] Patt YZ, Hassan MM, Aguayo A, Nooka AK, Lozano RD, Curley SA, Vauthey JN, Ellis LM, Schnirer II, Wolff RA, Charnsangavej C, Brown TD. Oral capecitabine for the treatment of hepatocellular carcinoma, cholangiocarcinoma, and gallbladder carcinoma. Cancer. 2004 Aug 1;101(3):578-86. doi: 10.1002/cncr.20368. PMID 15274071
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Van Cutsem E, Twelves C, Cassidy J, Allman D, Bajetta E, Boyer M, Bugat R, Findlay M, Frings S, Jahn M, McKendrick J, Osterwalder B, Perez-Manga G, Rosso R, Rougier P, Schmiegel WH, Seitz JF, Thompson P, Vieitez JM, Weitzel C, Harper P; Xeloda Colorectal Cancer Study Group. Oral capecitabine compared with intravenous fluorouracil plus leucovorin in patients with metastatic colorectal cancer: results of a large phase III study. J Clin Oncol. 2001 Nov 1;19(21):4097-106. doi: 10.1200/JCO.2001.19.21.4097. PMID 11689577
- [Background] Twelves CJ. Xeloda in Adjuvant Colon Cancer Therapy (X-ACT) trial: overview of efficacy, safety, and cost-effectiveness. Clin Colorectal Cancer. 2006 Nov;6(4):278-87. doi: 10.3816/CCC.2006.n.046. PMID 17241512
- [Background] Twelves C, Wong A, Nowacki MP, Abt M, Burris H 3rd, Carrato A, Cassidy J, Cervantes A, Fagerberg J, Georgoulias V, Husseini F, Jodrell D, Koralewski P, Kroning H, Maroun J, Marschner N, McKendrick J, Pawlicki M, Rosso R, Schuller J, Seitz JF, Stabuc B, Tujakowski J, Van Hazel G, Zaluski J, Scheithauer W. Capecitabine as adjuvant treatment for stage III colon cancer. N Engl J Med. 2005 Jun 30;352(26):2696-704. doi: 10.1056/NEJMoa043116. PMID 15987918
- [Background] Stockler M, S.T., Grimison P, et al, A randomized trial of capecitabine (C) given intermittently (IC) rather than continuously (CC) compared to classical CMF as first-line chemotherapy for advanced breast cancer (ABC). J Clin Oncol, 2007. 25(18S; June 20 suppl). Abstract 1031.
- [Background] Soto C, T.L., Reyes S, et al., Capecitabine (X) and taxanes in patients (pts) with anthracycline-pretreated metastatic breast cancer (MBC): sequential vs. combined therapy results from a MOSG randomized phase III trial. J Clin Oncol., 2006. 24(18S; June 20 suppl). Abstract 570.
- [Background] O'shaughnessy J, B.J., A retrospective evaluation of the impact of dose reduction in patients treated with Xeloda (capecitabine). Proc Am Soc Clin Oncol, 2000. 19: 104a. Abstract 400.